CLINICAL TRIAL: NCT06209567
Title: An Investigator-Initiated Study to Evaluate PSMA Expression in Patients With High-Grade Gliomas or Brain Metastases With 68Ga-PSMA-11 PET
Brief Title: A Study of 68Ga-PSMA-11 PET Scans in People With Brain Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-382
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: High-grade Glioma; Brain Metastases; Brain Metastases, Adult
Keywords: 68Ga-PSMA-11; High-grade Glioma; Brain Metastases; 23-382; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants with high-grade glioma (Experimental): Participants with newly diagnosed or recurrent high-grade glioma/HGG or brain metastases
  Interventions: Diagnostic Test: 68Ga-PSMA-11 PET Scans

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA-11 PET Scans — Participants will be injected intravenously with 68Ga-PSMA-11 via intravenous catheter. PET scans will first be interpreted without information on the results of other imaging modalities. Following the blinded read of the 68Ga-PSMA-11 PET scans, all recorded findings will be correlated with the results of CE CT and MR studies and 18F-FDG PET/CT or PET/MR performed as part of standard clinical care.

SUMMARY:
The purpose of this study is to find out whether 68Ga-PSMA-11 PET/CT is effective in assessing tumor uptake (tumor activity seen in cancerous tissue) in participants with high-grade glioma/HGG or brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign (or their legally acceptable representative (LAR) must sign) a written informed consent document
* Adults ≥ 18 years old
* Suspicion for or histologically or cytologically confirmed and previously treated HGG or brain metastases from a primary extracranial malignancy
* Lesion size ≥ 1 cm (for the lesion to be biopsied)
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Planned to undergo biopsy/resection of brain lesion

Exclusion Criteria:

* Inability to undergo a PET scan (e.g., claustrophobia or noncompatible implant in case PET/MR is performed)
* Pregnant or nursing female. All women of childbearing potential must have a documented negative serum or urine pregnancy test <1 week before study.
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiacarrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with severe allergy to both iodinated and gadolinium contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Assess range of tumor uptake of 68Ga-PSMA-11 in participants | up to 12 months
  Intensity and range of tumor uptake of 68Ga-PSMA-11 will be described using the SUVmean and SUVmax

CONTACTS AND LOCATIONS:
Overall Officials: Anton Nosov, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org